CLINICAL TRIAL: NCT00542321
Title: Multi-site Randomized Clinical Trial of Horizontal Positioning to Prevent and Treat Pulmonary Complications in Mechanically Ventilated Critically Ill Patients
Brief Title: Pilot Study of Lateral Rotation Interventions for Efficacy and Safety in ICU Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Society of Critical Care Medicine (Other)
Responsible Party: Principal Investigator, Sandra K. Hanneman, Professor - UT School of Nursing, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMCSCCMAACN
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Pneumonia, Ventilator Associated
Keywords: lateral rotation; kinetic therapy; mechanical ventilation; pulmonary complications
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinetic Therapy Bed (Experimental): Kinetic Therapy Bed: Continuous automated turning to 45 degrees with head of the bed elevated 30 degrees or more for up to 7 continuous days
  Interventions: Device: kinetic therapy bed
- Manual Turn (Active Comparator): Manual Turn: lateral rotation every 2 hours from back to left to back to right to back, with >/= 45 degree lateral rotation angle and 30 degree head of bed elevation
  Interventions: Other: Manual turn

INTERVENTIONS:
Other: Manual turn — Manual turn from side to back to side every 2 hours by nurses while patient receiving mechanical ventilation
  Other Names: Lateral rotation
  Arms: Manual Turn
Device: kinetic therapy bed — Continuous, automated turning to a maximum of 45 degrees in the lateral positions while the patient is receiving mechanical ventilation
  Other Names: CLRT (continuous lateral rotation therapy); KT (kinetic therapy)
  Arms: Kinetic Therapy Bed

SUMMARY:
Intensive care unit (ICU) patients on respirators are at high risk for preventable pulmonary complications (PPC). Turning these patients from side to side may reduce PPC, but carries the burden of decreases in blood pressure and oxygenation. The investigators hypothesize that there will be no difference in PPC or adverse events when ICU patients on respirators are turned by nurses or by an automated turning bed.

DETAILED DESCRIPTION:
The purpose of this pilot study is to test the feasibility of two turning protocols and study procedures for a multi-site randomized clinical trial to evaluate efficacy and safety of horizontal positioning interventions to reduce pulmonary complications in mechanically ventilated critically ill adult patients. The hypothesis of the randomized controlled trial (RCT) is no difference in pulmonary complications between manual, 2-hourly lateral rotation to > 45 degrees (control), and continuous automated turning to 45 degrees (experimental) groups.

ELIGIBILITY:
Inclusion Criteria:

* receiving mechanical ventilation
* ability to place on study protocol within 8 hours of intubation

Exclusion Criteria:

* pulmonary mass, pneumothorax, hemothorax, pleural effusion, or other source of compression atelectasis at time of assessment for eligibility
* systolic blood pressure < 90 mmHg with vasopressor support
* orthopedic injuries requiring limited or complete immobilization
* head injury requiring intracranial pressure monitoring
* unstable spinal injuries
* rib fractures
* body weight > 350 lbs
* intubation within the previous 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K. Hanneman, PhD, RN, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Background] Padhye NS, Cron SG, Gusick GM, Hamlin SK, Hanneman SK. Randomization for clinical research: an easy-to-use spreadsheet method. Res Nurs Health. 2009 Oct;32(5):561-6. doi: 10.1002/nur.20341. PMID 19606450
- [Background] Hamlin SK, Hanneman SK, Wachtel S, Gusick G. Adverse hemodynamic effects of lateral rotation during mechanical ventilation. Dimens Crit Care Nurs. 2008 Mar-Apr;27(2):54-61. doi: 10.1097/01.dcc.0000311593.87097.6a. PMID 18510182
- [Background] Padhye NS, Hamlin S, Brazdeikis A, Hanneman SK. Cardiovascular impact of manual and automated turns in ICU. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:1844-7. doi: 10.1109/IEMBS.2009.5332599. PMID 19963521
- [Background] Hanneman SK, Gusick GM, Hamlin SK, Wachtel SJ, Cron SG, Jones DJ, Oldham SA. Manual vs automated lateral rotation to reduce preventable pulmonary complications in ventilator patients. Am J Crit Care. 2015 Jan;24(1):24-32. doi: 10.4037/ajcc2015171. PMID 25554551
- [Background] Hamlin SK, Hanneman SK, Padhye NS, Lodato RF. Hemodynamic changes with manual and automated lateral turning in patients receiving mechanical ventilation. Am J Crit Care. 2015 Mar;24(2):131-40. doi: 10.4037/ajcc2015782. PMID 25727273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period spanned 8.6 months (between 09/28/07 - 04/30/07 and 05/01/09 - 08/31/09) and was done in 2 ICUs of 2 tertiary hospitals. Recruitment efforts were intermittent due to staffing resources and reconfiguration and testing of automated turn bed angle sensor.
Pre-assignment Details: Not applicable. All enrolled patients assigned to group.
Groups:
- Manual Turn: Manual Turn: lateral rotation every 2 hours from back to left to back to right to back, with >/= 45 degree lateral rotation angle and 30 degree head of bed elevation for up to 7 consecutive days
Period: Overall Study
Arm/Group | Kinetic Therapy Bed | Manual Turn
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kinetic Therapy Bed | Manual Turn | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11.4) | 54.3 (12.2) | 56.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Vasopressor Use [Number; unit: Participant] — Use of continuous intravenous infusion of any vasopressor during study period
  Participant
    Presence | 3 | 3 | 6
    Absence | 5 | 5 | 10
COPD Diagnosis [Number; unit: Participant] — Diagnosis of chronic obstructive pulmonary disease (COPD) in medical record
  Participant
    Yes | 0 | 4 | 4
    No | 8 | 4 | 12
Surgery [Number; unit: Participant]
  Yes | 3 | 2 | 5
  No | 5 | 6 | 11
APACHE II [Mean (Standard Deviation); unit: Scores on a scale] — Score on the Acute Physiology and Chronic Health Evaluation (APACHE) II (acuity of illness)instrument. Score ranges from 0 to 71, with higher score indicating greater severity of illness and risk for mortality.
  Scores on a scale | 24 (5) | 27 (9) | 25 (6.7)
FIO2 [Mean (Standard Deviation); unit: Fraction] — Fraction of inspired oxygen (FIO2) from APACHE II assessment (highest FIO2 within 24 hours of ICU admission)
  Fraction | 0.73 (0.25) | 0.77 (0.28) | 0.75 (0.26)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pulmonary Complications.
Description: Number of participants who did not have preventable pulmonary complications (PPC) on pre-study chest radiograph (CXR) and developed PPC during the study period. Pearson Chi-Square test used to test significance of difference between turning groups.
Time Frame: Participants were followed for the duration of ICU stay, an average of 10 days.
Population: Intention to treat; all 8 patients enrolled in kinetic therapy bed turn and 7 of 8 patients enrolled in manual turn (1 died before protocol initiated)
Measure: Number; unit: participants
Arm/Group | Kinetic Therapy Bed | Manual Turn
Number analyzed (Participants) | 8 | 7
participants | 1 | 1
Statistical Analysis 1: Comparison: Kinetic Therapy Bed vs Manual Turn; Pearson Chi-Square Test for difference between groups; Test type: Superiority or Other; p = 1.00, Fisher Exact; Chi-Square = 0.750, df = 1; difference between proportions = .5

2. Secondary Outcome: Mechanical Ventilation Duration.
Description: Days on mechanical ventilation, from initiation to withdrawal of mechanical ventilation
Time Frame: Participants were followed for the duration of mechanical ventilation, an average of 5.5 days.
Population: All 8 patients enrolled in kinetic therapy bed group and 7 of 8 patients enrolled in manual turn group (1 death before study protocol initiated)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Kinetic Therapy Bed | Manual Turn
Number analyzed (Participants) | 8 | 7
Days | 5.97 (4.99) | 5.21 (4.29)
Statistical Analysis 1: Comparison: Kinetic Therapy Bed vs Manual Turn; There will be no difference in duration of mechanical ventilation between groups; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney) — Alpha = .05; Rank sums = 52

3. Secondary Outcome: ICU Length of Stay.
Description: Time in days from study ICU admission to study ICU discharge or death
Time Frame: Participants were followed for the duration of ICU stay, an average of 10 days.
Population: All 8 patients enrolled in kinetic therapy bed group and 7 of 8 patients enrolled in manual turn group (1 patient enrolled but died before started on protocol)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Kinetic Therapy Bed | Manual Turn
Number analyzed (Participants) | 8 | 7
Days | 11.1 [5.4 to 23.4] | 8.2 [3.6 to 14.9]
Statistical Analysis 1: Comparison: Kinetic Therapy Bed vs Manual Turn; Test type: Superiority or Other; p = 0.451, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: ICU All-cause Mortality.
Description: Death from any reason between admission and discharge from study ICU
Time Frame: Participants were followed for the duration of ICU stay, an average of 10 days.
Population: All 8 patients enrolled in the kinetic therapy bed group and 7 of the 8 patients enrolled in the manual turn group (1 patient died before start of study protocol)
Measure: Number; unit: participants
Arm/Group | Kinetic Therapy Bed | Manual Turn
Number analyzed (Participants) | 8 | 7
participants | 2 | 2
Statistical Analysis 1: Comparison: Kinetic Therapy Bed vs Manual Turn; Test type: Superiority or Other; p = 1.0, Fisher Exact; probability = 0.430

5. Secondary Outcome: Turning-related Events
Description: Non-serious adverse events that occurred during the time of rotation in the kinetic therapy bed group and during lateral rotation to right or left position in the manual turn group
Time Frame: Participants were followed for the duration of time on protocol, an average of 3.5 days.
Population: All 8 patients enrolled in the kinetic therapy bed group and 7 of the 8 patients enrolled in the manual turn group (1 patient died after enrollment but before protocol could be initiated)
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Kinetic Therapy Bed | Manual Turn
Number analyzed (Participants) | 8 | 7
Events | 138 (131) | 125 (87)
Statistical Analysis 1: Comparison: Kinetic Therapy Bed vs Manual Turn; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney); Rank sums = 56

ADVERSE EVENTS:
Time Frame: Time on protocol (7 days or less)
Arm/Group | Kinetic Therapy Bed | Manual Turn
Serious Adverse Events (participants affected / at risk) | 4/8 | 3/7
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kinetic Therapy Bed (N=8) | Manual Turn (N=7)
Death (General disorders) | 1 (1) | 0 (0) — Planned death with withdrawal of life support
Dysrhythmia (Cardiac disorders) | 1 (2) | 1 (1) — Includes tachycardia, atrial fibrillation, and supraventricular tachycardia
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Marked decrease in peripheral oxygen saturation
Inadvertent extubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient self-extubation
Hypertension (General disorders) | 3 (3) | 0 (0) — Increase in mean arterial blood pressure > 20 mm Hg sustained for 5 minutes or more
Hypotension (General disorders) | 0 (0) | 1 (1) — Decrease in mean arterial pressure > 20 mm Hg sustained for 5 minutes or more
Ventilator Disconnection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Inadvertent disconnection of ventilator from endotracheal tube
Ventilator malfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kinetic Therapy Bed (N=8) | Manual Turn (N=7)
Discomfort:Psychologic (Psychiatric disorders) | 8 (227) | 7 (300) — Includes such observations as anxiety, apprehension, confusion, disorientation, agitation, change in Richmond Agitation Sedation Scale score
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 8 (525) | 7 (213) — Includes such observations and patient complaints as cough, shortness of breath, tachypnea, SpO2 changes </= 4%, tension on the endotracheal tube/ventilator tubing, patient-ventilator dysynchrony, bronchial secretions, and cuff leak
Hemodynamic (Vascular disorders) | 8 (237) | 6 (243) — Includes such observations as change in systolic blood pressure </= 19 mmHg and/or heart rate </= 29 beats/min, and dysrhythmias
Discomfort:Physiologic (General disorders) | 8 (59) | 6 (74) — Includes such observations or patient complaints as faintness, dizziness, fear of falling, and pain
Miscellaneous (General disorders) | 6 (48) | 4 (36) — Includes such observations as rectal thermometry probe/sensor displacement, neuromuscular manifestations, and bleeding
Skin (Skin and subcutaneous tissue disorders) | 1 (4) | 3 (8) — Includes pressure ulcers and skin lesions other than pressure ulcers

LIMITATIONS AND CAVEATS:
Reliance on chest X-ray interpretation only for detection of preventable pulmonary complications; small pilot study; kinetic therapy bed turn angle was less than 45 degrees

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No